CLINICAL TRIAL: NCT03131024
Title: The Effects of Short-term Exercise or Caloric Restriction on Anthracycline Chemotherapy-related Treatment Toxicity
Brief Title: Caloric Restriction and Exercise for Protection From Anthracycline Toxic Effects
Acronym: CREATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HREBA.CC-17-0129
Record Dates: First submitted 2017-04-21; First posted 2017-04-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer Female
Keywords: anthracyclines
MeSH Terms: interventions — Caloric Restriction; Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercise (Experimental): The exercise arm includes a single bout of supervised treadmill walking scheduled such that it would end approximately 24 hours prior to each of the participant's scheduled anthracycline treatment time.
  Interventions: Other: Aerobic exercise
- 50% caloric restriction (Experimental): The caloric restriction arm will restrict their total caloric intake by 50% for 48 hours prior to each anthracycline treatment.
  Interventions: Dietary Supplement: 50% caloric restriction
- Usual care (No Intervention): The usual care arm will be asked to maintain their typical exercise and diet throughout treatment.

INTERVENTIONS:
Dietary Supplement: 50% caloric restriction — Meals mimicking participant dietary preferences and matching North American macronutrient guidelines will be provided consisting of 50% of total caloric intake for 48 hours
  Arms: 50% caloric restriction
Other: Aerobic exercise — The supervised exercise session will consist of a 10-minute warm-up, 30 minutes performed at 70-75% of heart rate reserve, which corresponds to a vigorous intensity, followed by a 5-minute cool-down
  Arms: Aerobic exercise

SUMMARY:
Doxorubicin and epirubicin are part of the class of chemotherapy agents called anthracyclines that are commonly used to treat breast cancer. Although these treatments work well against the tumor, they are known to cause damage to the heart muscle, resulting in diminished heart function that can be permanent, and may also damage the blood vessels and skeletal muscles. The purpose of this study is to determine whether short-term application of these interventions with specific timing relative to the receipt of each treatment can prevent the negative effects of anthracycline treatment on the heart, aorta (largest artery leaving the heart), and skeletal muscle, and reduce treatment symptoms. Fifty-six early stage breast cancer patients who will receive anthracycline treatment will be randomly assigned to 1 of 3 groups who will: 1) perform a single 30-minute aerobic exercise session 24 hours prior to each treatment; 2) eat a diet consisting of 50% less calories for 48 hours prior to each treatment; or 3) receive usual cancer care. Magnetic resonance imaging (MRI) will be used to precisely measure the function of the heart, aorta, and the lower leg skeletal muscle at rest, and again during exercise to allow detection of more subtle signs of damage. We will also measure exercise capacity (i.e. aerobic fitness), microscopic damage to the heart muscle cells, a marker released into the blood in response to anthracycline-related heart damage, tumor size in patients receiving chemotherapy before surgery, quality of life and fatigue. These measures will be performed before treatment, at the end of treatment and 1 year later.

DETAILED DESCRIPTION:
Research Question: Is there a practical, widely available, non-pharmacological intervention that can be used to reduce the detrimental effects of anthracycline treatment to improve breast cancer patient cardiovascular health, well-being?

Primary Hypothesis: short-term application of aerobic exercise or caloric restriction prior to anthracycline chemotherapy treatments for breast cancer will reduce the detrimental effects of anthracyclines on heart, vessels and skeletal muscle.

Exploratory Hypothesis: these interventions will enhance the anticancer effects of anthracyclines and/or reduce the detrimental effects of anthracyclines on health-related quality of life.

Primary Study Aims: to investigate the effect of a single aerobic exercise session performed 24 hours prior to anthracycline treatment and the effect of 50% caloric restriction for 48 hours prior to anthracycline treatment relative to usual care control. Specifically, we will measure the intervention effects on:

I) Cardiac structure and function: 1) circulating NT-proBNP (interventions will mitigate unwanted increase in this prognostic marker of development of later cardiotoxicity); 2) left ventricular ejection fraction reserve (interventions will mitigate unwanted reduction in ability to augment heart function with exercise challenge) and 3) cardiac T1 mapping (interventions will mitigate unwanted increase in this marker of formation of myocardial fibrosis)

II) Vascular Function: 1) Aortic distensibility (rest) (interventions will mitigate unwanted increase in vascular stiffness)

III) Skeletal Muscle Structure and Function: 1) skeletal muscle oxygen consumption 2) skeletal muscle oxygen extraction (interventions will mitigate unwanted loss of oxygen consumption, extraction at peak exercise and in recovery) and 3) skeletal muscle mass and quality (interventions will mitigrate unwanted loss of skeletal muscle mass and quality).

Exploratory Study Aims: to investigate the effects of these interventions relative to the control group on: 1) tumor size at end of treatment in neoadjuvant patients (interventions will reduce tumor size) and 2) quality of life and fatigue at end of treatment and one year after treatment (interventions will improve quality of life and fatigue) and 3) long-term clinical cardiac and cancer outcomes.

Design and Recruitment:

This study will be a three-arm randomized control trial of fifty-six early stage breast cancer patients receiving adjuvant or neoadjuvant anthracycline-containing chemotherapy treatment. Following completion of the baseline assessment, participants will randomized to one of three groups who will: 1) complete a supervised vigorous intensity aerobic exercise session 24 hours prior to each anthracycline treatment; 2) restrict their caloric intake by 50% for 48 hours prior to each treatment; or 3) control condition receiving oncological usual care only. Participants will be recruited via oncologist referral from the Cross Cancer Institute.

Sample Size Determination:

Cardiac MRI is extremely reproducible and thus sensitive to detecting change in ejection fraction. It has been previously demonstrated that n=15 patients are required to detect a 3 percentage point change of resting ejection fraction with cardiac MRI, an 85% reduction in sample size required to detect the same change using echocardiography. Using a n=15 sample size per group for a three-arm, three-repeated measures design, there is >90% power to detect a medium effect size at p=0.05 (G*Power Version 3.0.10, F-test with repeated measures and a within-between factor design). The primary outcome in the current study, ejection fraction reserve (peak ejection fraction minus resting ejection fraction) is expected to be more sensitive than resting ejection fraction and therefore this sample size is expected to detect a difference between the intervention groups and the control group. We will enrol n=56 total (n=18-19 per group) to allow for a 20% rate for dropout, death, and technical difficulties.

Statistical Methods:

Given the longitudinal study design with data collected at 3 time points for each subject, a linear mixed model analysis that includes both fixed and random effects, with an intention to treat approach will be used. The repeated measures on a single subject result in correlated outcome data, and the random effects allow this correlation to be explicitly modeled. An additional advantage is that it allows for missing data on a subject without deleting all the data for that subject. The model also allows for covariates to be tested and can include time varying covariates (e.g. treatments received post anthracyclines). One assumption of mixed models is that the residuals from the model are normally distributed. Pilot data indicates that this assumption will hold for this study. If that is not the case, a Generalized Linear Mixed Model analysis, which can fit other distributions, will be used. All analyses will be performed using SPSS 24.0.

An interim analysis of resting ejection fraction only (standard parameter used to monitor cardiotoxicity within oncology practice) will be completed by a paid statistician not associated with the study. Resting ejection fraction will be compared between groups after completion of the end of treatment assessment for the first thirty participants. A second interim analysis will be performed upon suggestion by the statistician.

ELIGIBILITY:
Inclusion Criteria:

* age 18+
* Female
* stage I-IIIC breast cancer
* scheduled to receive an anthracycline-containing chemotherapy protocol
* able to read and communicate in English
* willing and able to adhere to either intervention

Exclusion Criteria:

* contraindications to MRI (e.g. pacemakers, metal implants)
* contraindications to maximal exercise testing
* pregnant
* have orthopedic limitations to sustained exercise on all potential modes (treadmill, elliptical, bike)
* have a body mass index <19 kg/m2
* history of eating disorder (self- or oncologist-reported)
* diabetes
* severe food allergies or restrictions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction reserve (peak exercise - rest) | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Cine steady-state free precession 2- and 4- chamber images will be taken at rest and at peak exercise using a resisted stepping device with a 3 T MRI scanner

SECONDARY OUTCOMES:
Change in NT-proBNP | 3-14 days before first anthracycline treatment, 24 hours after 1st and last anthracycline treatments, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  NT-proBNP will be analyzed in serum using electrochemiluminescence sandwich immunoassays
Change in aortic distensibility | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Transverse cine images of the ascending and descending aorta will be taken with a 3 T MRI scanner
Change in skeletal muscle oxygen extraction reserve (peak exercise - rest) | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Susceptometry-based oximetry using deoxyhemoglobin as an intrinsic contrast agent measured at rest and at peak exercise using a resisted plantar flexion device with a 3 T MRI scanner
Change in skeletal muscle oxygen consumption reserve (peak exercise - rest) | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Susceptometry-based oximetry using deoxyhemoglobin as an intrinsic contrast agent, coupled with phase contrast imaging for simultaneous measurement of lower leg blood flow, will together yield oxygen consumption, which will be measured at rest and at peak exercise using a resisted plantar flexion device with a 3 T MRI scanner
Change in resting LV strain | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Strain will be measured from cine steady-state free precession 2- and 4- chamber images will be taken at rest with a 3 T MRI scanner
Change in peak exercise LV strain | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Strain will be measured from cine steady-state free precession 2- and 4- chamber images will be taken at peak exercise using a resisted stepping device with a 3 T MRI scanner
Change in cardiac T1 | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  T1 mapping will performed in a mid-ventricular short-axis slice using saturation recovery single-shot acquisition (SASHA) pulse and Modified Look-Locker inversion recovery (MOLLI) sequencing
Change in peak LVEF | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Cine steady-state free precession 2- and 4- chamber images will be taken at peak exercise using a resisted stepping device with a 3 T MRI scanner
Patient-reported treatment symptoms | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  The Rotterdam Symptom Checklist will be used to rate the prevalence and severity of treatment symptoms
Change in cardiac output | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Cine steady-state free precession will be taken at rest and peak exercise to quantify volumes and will be multiplied by heart rate to determine cardiac output
Change in LV volumes | Cine steady-state free precession will be taken at rest and peak exercise to quantify volumes and will be multiplied by heart rate to determine cardiac output
  Cine steady-state free precession will be taken at rest and peak exercise to quantify volumes
Change in resting LVEF | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Cine steady-state free precession 2- and 4- chamber images will be taken at rest
Change in LV mass | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Mass will be measured using MRI
Change in thigh skeletal muscle mass and quality | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Skeletal muscle mass of the thigh will be measured using Dixon fat-water separation imaging method that yields separated water and fat images to quantify skeletal muscle and adipose tissue.
Change in peak oxygen consumption | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Peak oxygen consumption will measured using a maximal cardiopulmonary exercise test

OTHER OUTCOMES:
Health-related quality of life and fatigue | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment, one year after initiation of anthracycline treatment
  Health-related quality of life will be measured by the Functional Assessment of Cancer Therapy - Fatigue (FACT-F) questionnaire.
Change in clinical tumor size | Anytime prior to inititiation of chemotherapy, and within 1 month of completion of chemotherapy or as otherwise clinically indicated
  Clinical tumor size will be assessed using ultrasound in participants receiving neoadjuvant chemotherapy only
Combined clinical end-point | 1 and 5 years after completion of treatment
  cancer recurrence, cardiac events, hospitalizations, and mortality will be extracted from clinical records and combined into a clinical end-point
Change in circulating markers of oxidative stress/antioxidants | 3-14 days before first anthracycline treatment, 2-3 weeks after completion of anthracycline treatment
  ELISA assays will be used to measure circulating markers of oxidative stress such as MDA and antioxidants such as Mn-SOD. Due to rapid development of these types of assays, samples will be frozen and will be run in batch analysis at the end of the study such that the most modern assays can be used.

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Kirkham, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirkham AA, Paterson DI, Prado CM, Mackey JR, Courneya KS, Pituskin E, Thompson RB. Rationale and design of the Caloric Restriction and Exercise protection from Anthracycline Toxic Effects (CREATE) study: a 3-arm parallel group phase II randomized controlled trial in early breast cancer. BMC Cancer. 2018 Sep 3;18(1):864. doi: 10.1186/s12885-018-4778-7. PMID 30176834